CLINICAL TRIAL: NCT05263375
Title: TVMR With the Innovalve System Trial - Pilot Study in Belgium
Brief Title: TVMR With the Innovalve System Trial - TWIST-BE TWIST-PILOT-BE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stdy never submitted to any regulatory body or never initiated
Sponsor: Innovalve Bio Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INVL21-02-BE
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MV replacement with Innovalve TMVR system (Experimental): MV replacement with Innovalve TMVR system
  Interventions: Device: Innovalve TMVR system

INTERVENTIONS:
Device: Innovalve TMVR system — Innovalve TMVR system

SUMMARY:
Study to evaluate the safety and performance of the Innovalve mitral valve replacement system

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant, symptomatic mitral regurgitation
* High risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Patient is inoperable
* EF <30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with implant or delivery related serious adverse events at 30 days | 30 days
  Number of patients with implant or delivery related serious adverse events at 30 days